CLINICAL TRIAL: NCT05552209
Title: Assessment of the Safety and Performance of Elbow Supports in the Context of Epicondylitis or a Return to Sport After Sprain
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Decathlon SE (Industry)
Collaborators: EFOR, France (Industry)
Responsible Party: Sponsor
Other Study IDs: elbowMID500-STRAP
Record Dates: First submitted 2022-09-13; First posted 2022-09-23 (Actual); Last update posted 2023-01-17 (Actual); Status verified 2023-01

CONDITIONS: Epicondylitis; Elbow Sprain

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Orthosis group 1: Use of Elbow Mid 500 device during sport practice
  Interventions: Device: Elbow MID 500
- Control group 1: Control group of the Elbow Mid 500 group - no medical device used during sport practice
  Interventions: Other: Control group Elbow MID 500
- Orthosis group 2: Use of Elbow Strap device during sport practice
  Interventions: Device: Elbow STRAP
- Control group 2: Control group of the Elbow Strap group - no medical device used during sport practice
  Interventions: Other: Control group Elbow STRAP

INTERVENTIONS:
Device: Elbow MID 500 — 15 patients will be included in this group and will used the medical device Elbow MID 500 during sport practice (at least 2 sport sessions per week), for 6 weeks.
  Groups: Orthosis group 1
Other: Control group Elbow MID 500 — 15 patients will be included in this control group and will performed their sport sessions as usual (without the medical device Elbow MID 500), for at least 2 sport sessions per week during 6 weeks.
  Groups: Control group 1
Device: Elbow STRAP — 15 patients will be included in this group and will used the medical device Elbow STRAP during sport practice (at least 2 sport sessions per week), for 6 weeks.
  Groups: Orthosis group 2
Other: Control group Elbow STRAP — 15 patients will be included in this control group and will performed their sport sessions as usual (without the medical device Elbow STRAP), for at least 2 sport sessions per week during 6 weeks.
  Groups: Control group 2

SUMMARY:
Decathlon has developed elbowMID500 and elbowSTRAP products which are medical devices that must be positioned around the elbow during sport practice, in order to limit symptoms related to epicondylitis or previous sprains (elbowMID500 only).

The objective of this multicentre study is to collect data on the related clinical complications and clinical outcomes of market-approved Decathlon elbowMID500 and elbowSTRAP products to demonstrate safety and performance of these devices in a real-world setting.

Outcome data collected from this study will provide the basis for Post-Market Surveillance (PMS) reporting, Clinical Study Report (CSR), Clinical Evaluation Report (CER) on Decathlon elbowMID500 and elbowSTRAP devices and support peer-reviewed publications on products performance and safety.

ELIGIBILITY:
Inclusion Criteria:

* Subject is aged ≥ 18 years old
* Subject has an acute epicondylitis (stage 1 or 2) OR a recent mild elbow sprain
* Subject performs regular physical activity (minimum of 2 sessions of 10 minutes per week)
* The current condition of his/her elbow allows the subject to resume usual physical activity
* Subject has been informed and is willing to sign an informed consent form
* Subject is willing to comply with protocol requirements and return to the study center for all clinical evaluations and required follow-up (6 weeks)
* Subject is affiliated to the French social security regime

Exclusion Criteria:

* Subject has conditions that may interfere with his/her ability to understand protocol requirements, participate in scheduled visits, or provide his/her informed consent
* Subject has worn a support (elbow brace or articulated orthosis) in the last month during his/her sport practice
* Subject has resumed regular physical activity since his/her recent injury
* Subject has any medical condition that could impact the study at investigator's discretion
* Subject has a known hypersensitivity or allergy to the components of the device (polyamide, elastane, polyester, elastodiene) • Adult subject to legal protection measure

Ages: 18 Years to 99 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Subjects with acute epicondylitis (stage 1 or 2) or a recent mild elbow sprain whose current condition of their elbow allows them to pursue a usual physical activity.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-09-21 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
Functional score | Change from Baseline functionnal score at 6 weeks
  Comparison of the Japanese Elbow Assessment Score System (JOA elbow scale from 0=worst ouctome to 100=best outcome) between the baseline and last follow-up visit in each group (orthosis vs control), for each device model.

SECONDARY OUTCOMES:
Confidence level (confidence questionnaire related to physical activity) | Change from Baseline confidence level at 6 weeks
  Gap in the confidence level related to physical activity (scale from 0=worst outcome to 100=best outcome), between the baseline and last follow-up visit in each group (orthosis vs control), for each device model
Elbow pain | Change from Baseline elbow pain at 6 weeks
  Comparison of elbow pain, assessed through a Numerical Rating Scale (NRS) ranging from 0=best outcome to 10=worst outcome, between the groups (orthosis vs control), for each device model
Safety (adverse events) | 6 weeks of follow-up
  Comparison of adverse events rates between the groups (orthosis vs control), for each device model

CONTACTS AND LOCATIONS:
Overall Officials: Valérie WIECZOREK, Principal Investigator — Centre Hospitalier Universitaire de Lille
Locations (4):
- France (4):
  - Centre Hospitalier de Boulogne sur Mer, Boulogne-sur-Mer
  - Centre de rééducation et de balnéothérapie Kinés Faches, Faches-Thumesnil
  - Centre Hospitalier Universitaire de Lille, Lille
  - Cabinet de kinésithérapie du Belvédère, Paris

IPD SHARING:
Plan to Share IPD: No